CLINICAL TRIAL: NCT01338649
Title: Effects of Bright Light Treatment on Daytime Sleepiness and Nocturnal Sleep in Patients With Parkinson's Disease
Brief Title: Light Therapy Treatment in Parkinson's Disease Patients With Daytime Somnolence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Parkinson Foundation (Other)
Responsible Party: Principal Investigator, Aleksandar Videnovic, Assistant Professor of Neurology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Light Therapy in PD
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Parkinson's Disease; Sleep Disorder; Excessive Somnolence
Keywords: Parkinson's disease; Daytime somnolence; Sleepiness; Light therapy
MeSH Terms: conditions — Parkinson Disease; Sleep Wake Disorders; Disorders of Excessive Somnolence; Sleepiness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bright White (Active Comparator): Exposure to bright white light treatment.
  Interventions: Device: Bright Light Treatment (Sun Ray Sunbox SB-558)
- Dim red light (Placebo Comparator): Exposure to dim red light treatment.
  Interventions: Device: Dim red light (Sun Ray Sunbox SB-558)

INTERVENTIONS:
Device: Bright Light Treatment (Sun Ray Sunbox SB-558) — Bright Light Treatment (Sun Ray Sunbox SB-558) using light intensity of 10,000 lux, administered during two 1 hour periods during the day.
  Other Names: Sun Ray Sunbox SB-558
  Arms: Bright White
Device: Dim red light (Sun Ray Sunbox SB-558) — Dim red light box administered during two 1 hour periods during the day using
  Other Names: Sun Ray Sunbox SB-558
  Arms: Dim red light

SUMMARY:
Study objectives are to determine the efficacy, safety and tolerability of bright light treatment in Parkinson's Disease (PD) patients with daytime sleepiness. Thirty PD patients will be enrolled and equally randomized to bright light or dim-red light treatment. Objective (actigraphy) and subjective (sleep logs/scales) sleep measures will be collected through the baseline and intervention phases of the study. The primary outcome measure will be the change in the Epworth Sleepiness Scale (ESS) comparing the bright light treatment with dim-red light treatment. Secondary outcome measures will include the Multiple Sleep Latency Test (MSLT), global Pittsburgh Sleep Quality Index (PSQI) score, Parkinson's Disease Sleep Scale (PDSS) score, and actigraphy measures. A variety of exploratory analyses will examine the effects of bright light treatment on fatigue, depression, quality of life, cognition, and motor disability.

Hypothesis: Bright light exposure will diminish daytime sleepiness and improve night-time sleep in PD patients with daytime sleepiness.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD as defined by the United Kingdom Parkinson's Disease Society Brain Bank Criteria
2. Hoehn and Yahr stage of 2 to 4 in the "on" state
3. Excessive daytime sleepiness as defined by the Epworth Sleepiness Scale (ESS) score of greater than or equal to 12 points
4. Stable PD medication regimen for at least 4 weeks prior to study screening
5. Willing and able to give written informed consent

Exclusion Criteria:

1. Atypical parkinsonian syndromes
2. Significant sleep disordered breathing (defined as an apnea-hypopnea index >15 events/hr of sleep on screening PSG)
3. Significant periodic limb movement disorder (defined as a PLM arousal index>10 events/hr of sleep on screening PSG) and REM sleep behavior disorder (based on the presence of both clinical symptomatology as well as intermittent loss of REM atonia on screening PSG)
4. Cognitive impairment indicated by the mini-mental status examination (MMSE) score of less than 24
5. Presence of depression defined as the Beck Depression Inventory (BDI) score >14
6. Untreated hallucinations or psychosis (drug-induced or spontaneous)
7. Use of hypno-sedative drugs for sleep or stimulants during the daytime
8. Use of antidepressants unless the patient has been on a stable dose for at least three months
9. Visual abnormalities that may interfere with light therapy, such as significant cataracts, narrow angle glaucoma or blindness
10. Travel through 2 time zones within 90 days prior to study screening

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Videnovic, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Lees AJ, Blackburn NA, Campbell VL. The nighttime problems of Parkinson's disease. Clin Neuropharmacol. 1988 Dec;11(6):512-9. doi: 10.1097/00002826-198812000-00004. PMID 3233589
- [Background] Tandberg E, Larsen JP, Karlsen K. A community-based study of sleep disorders in patients with Parkinson's disease. Mov Disord. 1998 Nov;13(6):895-9. doi: 10.1002/mds.870130606. PMID 9827612
- [Background] Karlsen KH, Tandberg E, Arsland D, Larsen JP. Health related quality of life in Parkinson's disease: a prospective longitudinal study. J Neurol Neurosurg Psychiatry. 2000 Nov;69(5):584-9. doi: 10.1136/jnnp.69.5.584. PMID 11032608
- [Background] Scaravilli T, Gasparoli E, Rinaldi F, Polesello G, Bracco F. Health-related quality of life and sleep disorders in Parkinson's disease. Neurol Sci. 2003 Oct;24(3):209-10. doi: 10.1007/s10072-003-0134-y. PMID 14598091
- [Background] Meindorfner C, Korner Y, Moller JC, Stiasny-Kolster K, Oertel WH, Kruger HP. Driving in Parkinson's disease: mobility, accidents, and sudden onset of sleep at the wheel. Mov Disord. 2005 Jul;20(7):832-42. doi: 10.1002/mds.20412. PMID 15726539
- [Background] Factor SA, McAlarney T, Sanchez-Ramos JR, Weiner WJ. Sleep disorders and sleep effect in Parkinson's disease. Mov Disord. 1990;5(4):280-5. doi: 10.1002/mds.870050404. PMID 2259351
- [Background] Stocchi F, Barbato L, Nordera G, Berardelli A, Ruggieri S. Sleep disorders in Parkinson's disease. J Neurol. 1998 May;245 Suppl 1:S15-8. doi: 10.1007/pl00007731. PMID 9617717
- [Background] Paus S, Brecht HM, Koster J, Seeger G, Klockgether T, Wullner U. Sleep attacks, daytime sleepiness, and dopamine agonists in Parkinson's disease. Mov Disord. 2003 Jun;18(6):659-67. doi: 10.1002/mds.10417. PMID 12784269
- [Background] Rye DB, Bliwise DL, Dihenia B, Gurecki P. FAST TRACK: daytime sleepiness in Parkinson's disease. J Sleep Res. 2000 Mar;9(1):63-9. doi: 10.1046/j.1365-2869.2000.00201.x. PMID 10733691
- [Background] Lockley SW, Skene DJ, Arendt J, Tabandeh H, Bird AC, Defrance R. Relationship between melatonin rhythms and visual loss in the blind. J Clin Endocrinol Metab. 1997 Nov;82(11):3763-70. doi: 10.1210/jcem.82.11.4355. PMID 9360538
- [Background] Myers BL, Badia P. Changes in circadian rhythms and sleep quality with aging: mechanisms and interventions. Neurosci Biobehav Rev. 1995 Winter;19(4):553-71. doi: 10.1016/0149-7634(95)00018-6. PMID 8684716
- [Background] Moore RY, Eichler VB. Loss of a circadian adrenal corticosterone rhythm following suprachiasmatic lesions in the rat. Brain Res. 1972 Jul 13;42(1):201-6. doi: 10.1016/0006-8993(72)90054-6. No abstract available. PMID 5047187
- [Background] Dijk DJ, Lockley SW. Integration of human sleep-wake regulation and circadian rhythmicity. J Appl Physiol (1985). 2002 Feb;92(2):852-62. doi: 10.1152/japplphysiol.00924.2001. PMID 11796701
- [Background] Moore-Ede MC, Czeisler CA, Richardson GS. Circadian timekeeping in health and disease. Part 2. Clinical implications of circadian rhythmicity. N Engl J Med. 1983 Sep 1;309(9):530-6. doi: 10.1056/NEJM198309013090905. No abstract available. PMID 6348546
- [Background] Czeisler CA, Allan JS, Strogatz SH, Ronda JM, Sanchez R, Rios CD, Freitag WO, Richardson GS, Kronauer RE. Bright light resets the human circadian pacemaker independent of the timing of the sleep-wake cycle. Science. 1986 Aug 8;233(4764):667-71. doi: 10.1126/science.3726555.
- [Background] Wever RA, Polasek J, Wildgruber CM. Bright light affects human circadian rhythms. Pflugers Arch. 1983 Jan;396(1):85-7. doi: 10.1007/BF00584704. PMID 6835810
- [Background] Van Someren EJ, Riemersma RF, Swaab DF. Functional plasticity of the circadian timing system in old age: light exposure. Prog Brain Res. 2002;138:205-31. doi: 10.1016/S0079-6123(02)38080-4. No abstract available. PMID 12432772
- [Background] Shochat T, Martin J, Marler M, Ancoli-Israel S. Illumination levels in nursing home patients: effects on sleep and activity rhythms. J Sleep Res. 2000 Dec;9(4):373-9. doi: 10.1046/j.1365-2869.2000.00221.x. PMID 11386204
- [Background] Mishima K, Okawa M, Shimizu T, Hishikawa Y. Diminished melatonin secretion in the elderly caused by insufficient environmental illumination. J Clin Endocrinol Metab. 2001 Jan;86(1):129-34. doi: 10.1210/jcem.86.1.7097. PMID 11231989
- [Background] Klerman EB, Duffy JF, Dijk DJ, Czeisler CA. Circadian phase resetting in older people by ocular bright light exposure. J Investig Med. 2001 Jan;49(1):30-40. doi: 10.2310/6650.2001.34088. PMID 11217145
- [Background] Kobayashi R, Kohsaka M, Fukuda N, Sakakibara S, Honma H, Koyama T. Effects of morning bright light on sleep in healthy elderly women. Psychiatry Clin Neurosci. 1999 Apr;53(2):237-8. doi: 10.1046/j.1440-1819.1999.00486.x. PMID 10459698
- [Background] Kaida K, Takahashi M, Haratani T, Otsuka Y, Fukasawa K, Nakata A. Indoor exposure to natural bright light prevents afternoon sleepiness. Sleep. 2006 Apr;29(4):462-9. doi: 10.1093/sleep/29.4.462. PMID 16676779
- [Background] Phipps-Nelson J, Redman JR, Dijk DJ, Rajaratnam SM. Daytime exposure to bright light, as compared to dim light, decreases sleepiness and improves psychomotor vigilance performance. Sleep. 2003 Sep;26(6):695-700. doi: 10.1093/sleep/26.6.695. PMID 14572122
- [Background] Schindler SD, Graf A, Fischer P, Tolk A, Kasper S. Paranoid delusions and hallucinations and bright light therapy in Alzheimer's disease. Int J Geriatr Psychiatry. 2002 Nov;17(11):1071-2. doi: 10.1002/gps.497. PMID 12404657
- [Background] Fetveit A, Bjorvatn B. Bright-light treatment reduces actigraphic-measured daytime sleep in nursing home patients with dementia: a pilot study. Am J Geriatr Psychiatry. 2005 May;13(5):420-3. doi: 10.1176/appi.ajgp.13.5.420. PMID 15879592
- [Background] Dowling GA, Hubbard EM, Mastick J, Luxenberg JS, Burr RL, Van Someren EJ. Effect of morning bright light treatment for rest-activity disruption in institutionalized patients with severe Alzheimer's disease. Int Psychogeriatr. 2005 Jun;17(2):221-36. doi: 10.1017/s1041610205001584. PMID 16050432
- [Background] Ancoli-Israel S, Martin JL, Gehrman P, Shochat T, Corey-Bloom J, Marler M, Nolan S, Levi L. Effect of light on agitation in institutionalized patients with severe Alzheimer disease. Am J Geriatr Psychiatry. 2003 Mar-Apr;11(2):194-203. PMID 12611749
- [Background] Ancoli-Israel S, Gehrman P, Martin JL, Shochat T, Marler M, Corey-Bloom J, Levi L. Increased light exposure consolidates sleep and strengthens circadian rhythms in severe Alzheimer's disease patients. Behav Sleep Med. 2003;1(1):22-36. doi: 10.1207/S15402010BSM0101_4. PMID 15600135
- [Background] Dowling GA, Mastick J, Hubbard EM, Luxenberg JS, Burr RL. Effect of timed bright light treatment for rest-activity disruption in institutionalized patients with Alzheimer's disease. Int J Geriatr Psychiatry. 2005 Aug;20(8):738-43. doi: 10.1002/gps.1352. PMID 16035127
- [Background] Artemenko AR, Levin IaI. [The phototherapy of parkinsonism patients]. Zh Nevrol Psikhiatr Im S S Korsakova. 1996;96(3):63-6. Russian. PMID 8992840
- [Background] Reid KJ, Burgess HJ. Circadian rhythm sleep disorders. Prim Care. 2005 Jun;32(2):449-73. doi: 10.1016/j.pop.2005.02.002. PMID 15935195
- [Background] Kogan AO, Guilford PM. Side effects of short-term 10,000-lux light therapy. Am J Psychiatry. 1998 Feb;155(2):293-4. doi: 10.1176/ajp.155.2.293. PMID 9464216
- [Background] Dhawan V, Healy DG, Pal S, Chaudhuri KR. Sleep-related problems of Parkinson's disease. Age Ageing. 2006 May;35(3):220-8. doi: 10.1093/ageing/afj087. PMID 16638765
- [Background] Adler CH, Caviness JN, Hentz JG, Lind M, Tiede J. Randomized trial of modafinil for treating subjective daytime sleepiness in patients with Parkinson's disease. Mov Disord. 2003 Mar;18(3):287-293. doi: 10.1002/mds.10390. PMID 12621632
- [Derived] Videnovic A, Klerman EB, Wang W, Marconi A, Kuhta T, Zee PC. Timed Light Therapy for Sleep and Daytime Sleepiness Associated With Parkinson Disease: A Randomized Clinical Trial. JAMA Neurol. 2017 Apr 1;74(4):411-418. doi: 10.1001/jamaneurol.2016.5192. PMID 28241159

RESULTS

PARTICIPANT FLOW:
Groups:
- Bright White: Bright white light treatment group.
  Bright Light Treatment (Sun Ray Sunbox SB-558): Bright white light box using light intensity of 10,000 lux, administered during two 1 hour periods during the day.
- Dim Red Light: Dim red light control group.
  Dim red light (Sun Ray Sunbox SB-558): Dim red light box administered during two 1 hour periods during the day using
Period: Overall Study
Arm/Group | Bright White | Dim Red Light
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bright White | Dim Red Light | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (6.9) | 59.3 (11.3) | 63.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants] — number of participants
  participants
    United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in the Epworth Sleepiness Scale (ESS) Scores Comparing the Bright Light Exposure With Dim-red Light Exposure.
Description: ESS score range is 0-24; lower ESS scores indicate less daytime sleepiness; higher ESS scores indicate more severe sleepiness ESS will be taken and compared at screening and week 4 visits between the bright light exposure and dim-red light exposure groups.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Bright White | Dim Red Light
Number analyzed (Participants) | 13 | 14
score | 4.46 (2.54) | 1.77 (3)
Statistical Analysis 1: Comparison: Bright White vs Dim Red Light; Test type: Superiority or Other; p = 0.0211, t-test, 2 sided; t-test on two groups of differences

ADVERSE EVENTS:
Arm/Group | Bright White | Dim Red Light
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 2/13 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bright White (N=13) | Dim Red Light (N=14)
headache (Nervous system disorders) | 1 (1) | 0 (0)
sleepiness (Nervous system disorders) | 1 (1) | 0 (0)
itchy eyes (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No